CLINICAL TRIAL: NCT02096159
Title: Trimethoprim-sulfamethoxazole vs. Placebo After Hypospadias Repair: a Multicenter, Double-blind, Randomized Trial
Brief Title: Prophylactic Antibiotics or Placebo After Hypospadias Repair
Acronym: PROPHY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Earl Y Cheng, MD, Head, Division of Urology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LC/Uro-MF-01
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hypospadias
Keywords: Hypospadias; Anti-Bacterial Agents
MeSH Terms: conditions — Hypospadias | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotics (Experimental): trimethoprim-sulfamethoxazole oral suspension, 4 mg/kg (0.5 mL/kg) twice daily for 10 days
  Interventions: Drug: trimethoprim-sulfamethoxazole
- Placebo (Placebo Comparator): placebo oral suspension, 0.5 mL/kg twice daily for 10 days
  Interventions: Other: placebo

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole
  Arms: Antibiotics
Other: placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine if routine use of prophylactic (preventive) antibiotics after repair of mid-to-distal hypospadias is beneficial.

DETAILED DESCRIPTION:
Participants in this multicenter, double-blind study are randomized to receive trimethoprim-sulfamethoxazole or placebo for 10 days postoperatively. Short- and intermediate-term results will be published after participants complete 6 months and 5 years of follow-up, respectively.

ELIGIBILITY:
Inclusion Criteria:

* mid-to-distal shaft hypospadias
* single-stage hypospadias repair
* length of urethral repair (urethroplasty) less than or equal to 20 mm
* placement of an open-drainage urethral stent at the time of hypospadias repair, with intended duration of stenting for 5-10 days post-operatively

Exclusion Criteria:

* previous hypospadias repair
* prior adverse/allergic reaction or other contraindication to trimethoprim-sulfamethoxazole
* cross-reactivity of an existing medication with trimethoprim-sulfamethoxazole
* any patient condition with elevated risk of infection or adverse outcome from potential infection (e.g., HIV/AIDS, poorly controlled diabetes mellitus or other immunocompromising conditions, congenital heart disease)
* use of antibiotics within seven days prior to hypospadias repair
* foreskin reconstruction at the time of hypospadias repair
* prescription of oral antibiotics other than Study Medication at the time of hypospadias repair

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
postoperative infection | up to 30 days
  Urinary tract infection; cellulitis/wound infection
wound-healing complications | up to 5 years
  meatal stenosis; urethral stricture; urethrocutaneous fistula; dehiscence; urethral diverticulum

SECONDARY OUTCOMES:
adverse drug reaction | up to 14 days
C. difficile colitis | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Earl Y Cheng, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Mark A Faasse, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Faasse MA, Farhat WA, Rosoklija I, Shannon R, Odeh RI, Yoshiba GM, Zu'bi F, Balmert LC, Liu DB, Alyami FA, Beaumont JL, Erickson DL, Gong EM, Johnson EK, Judd S, Kaplan WE, Kaushal G, Koyle MA, Lindgren BW, Maizels M, Marcus CR, McCarter KL, Meyer T, Qureshi T, Saunders M, Thompson T, Yerkes EB, Cheng EY. Randomized trial of prophylactic antibiotics vs. placebo after midshaft-to-distal hypospadias repair: the PROPHY Study. J Pediatr Urol. 2022 Apr;18(2):171-177. doi: 10.1016/j.jpurol.2022.01.008. Epub 2022 Jan 25. PMID 35144885

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02096159/Prot_SAP_000.pdf